CLINICAL TRIAL: NCT03986112
Title: Ability of Carotid Sonography and Inferior Vena Cava Sonography for the Prediction of Post-induction Hypotension in Hypertensive Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2018-0064
Record Dates: First submitted 2019-06-12; First posted 2019-06-14 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: General Anesthesia
Keywords: carotid sonography; inferior vena cava sonography; hypertension; general anesthesia; predictive power
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hypertensive group: Evaluation of the ability of carotid sonography and inferior vena cava sonography for the post-induction hypotension in hypertensive patients undergoing general anesthesia
  Interventions: Biological: carotid sonography and inferior vena cava sonography

INTERVENTIONS:
Biological: carotid sonography and inferior vena cava sonography — Carotid and venous ultrasonography is performed in a comfortable state. Corrected blood flow after carotid ultrasound and carotid artery blood flow rate were measured. After inferior vena cava sonography, the collapsibility Index by measuring the largest and smallest diameter during the respiratory cycle will be obtained. Propofol 2 mg / kg is administered and remifentanil is maintained at 4.0 ng / mL using the Target Control System. Blood pressure and heart rate are measured at prior to induction, 1 minute after induction, immediately after intubation, and at 1, 3, 5, 7 and 10 minutes after intubation. Post-induction hypotension is considered as a decrease of 20% or more of baseline blood pressure or a mean arterial blood pressure of less than 60 mmHg. In the event of hypotension in accordance with the above definition, repeated administration of ephedrine 4 mg or phenylephrine 50 mcg is used.

SUMMARY:
Hypertensive patients have more hemodynamic instability during general anesthesia than do patients with NORMOTENSION. In this study, the investigators evaluated the usefulness of carotid ultrasound and inferior vena cervical ultrasound for predicting hypotension after induction of anesthesia in patients with hypertension.

DETAILED DESCRIPTION:
Carotid and venous ultrasonography is performed in a comfortable state. Corrected blood flow after carotid ultrasound and carotid artery blood flow rate were measured.

After inferior vena cava sonography, using the embedded software, the collapsibility Index by measuring the largest and smallest diameter during the respiratory cycle will be obtained.

After confirming baseline blood pressure and pulse rate, propofol 2 mg / kg is administered and remifentanil is maintained at 4.0 ng / mL using the Target Control System (TCI).

Following the administration of rocuronium 1.0-1.2 mg / kg, and 1 minute and 30 seconds after BIS 60 or less, endotracheal intubation is performed using video laryngoscope.

Blood pressure and heart rate are measured at prior to induction, 1 minute after the induction, immediately after intubation, and at 1, 3, 5, 7 and 10 minutes after intubation.

Post-induction hypotension after anesthesia induction is considered as a decrease of 20% or more of the pre-anesthesia blood pressure or a mean arterial blood pressure of less than 60 mmHg.

In the event of hypotension in accordance with the above definition, repeated administration of ephedrine 4 mg or phenylephrine 50 mcg is used.

ELIGIBILITY:
Inclusion Criteria:

* 1) 19-80 years old hypertensive patients with ASA class I-III
* 2) Scheduled surgery under general anesthesia

Exclusion Criteria:

* 1) Emergency operation
* 2) Reoperation
* 3) Patients with history of heart failure (unstable angina, congestive heart failure, coronary artery disease)
* 4) Patients under 40 % of Ejection faction
* 5) Patients with history of valvular heart failure
* 6) Patients with history of peripheral arterial occlusive disease
* 7) Patients with history of arrhythmia (specially AV nodal block), ventricular conduction problem
* 8) Pregnancy patients
* 9) Patients who cannot read the consent form (examples: Illiterate, foreigner)
* 10) Patients with history of uncontrolled psychiatric disease (PTSD, anxiety, depression)
* 11) Patients who withdraw the consent

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients aged 19 to 80 years who are scheduled to undergo surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Prediction power of the post-induction hypotension of carotid sonography and inferior vena cava sonography | Prior to induction
  To evaluate the ability of carotid sonography and inferior vena cava sonography for the post-induction hypotension in hypertensive patients undergoing general anesthesia, blood pressure was measured 8 times below time points.
Prediction power of the post-induction hypotension of carotid sonography and inferior vena cava sonography | 1 minute after anesthetic induction
  To evaluate the ability of carotid sonography and inferior vena cava sonography for the post-induction hypotension in hypertensive patients undergoing general anesthesia, blood pressure was measured 1 minute after anesthetic induction.
Prediction power of the post-induction hypotension of carotid sonography and inferior vena cava sonography | Immediately after intubation
  To evaluate the ability of carotid sonography and inferior vena cava sonography for the post-induction hypotension in hypertensive patients undergoing general anesthesia, blood pressure was measured Immediately after intubation.
Prediction power of the post-induction hypotension of carotid sonography and inferior vena cava sonography | 1 minute after tracheal intubation
  To evaluate the ability of carotid sonography and inferior vena cava sonography for the post-induction hypotension in hypertensive patients undergoing general anesthesia, blood pressure was measured 1 minute after tracheal intubation.
Prediction power of the post-induction hypotension of carotid sonography and inferior vena cava sonography | 3 minutes after tracheal intubation
  To evaluate the ability of carotid sonography and inferior vena cava sonography for the post-induction hypotension in hypertensive patients undergoing general anesthesia, blood pressure was measured 3 minutes after tracheal intubation.
Prediction power of the post-induction hypotension of carotid sonography and inferior vena cava sonography | 5 minutes after tracheal intubation
  To evaluate the ability of carotid sonography and inferior vena cava sonography for the post-induction hypotension in hypertensive patients undergoing general anesthesia, blood pressure was measured 5 minutes after tracheal intubation.
Prediction power of the post-induction hypotension of carotid sonography and inferior vena cava sonography | 7 minutes after tracheal intubation
  To evaluate the ability of carotid sonography and inferior vena cava sonography for the post-induction hypotension in hypertensive patients undergoing general anesthesia, blood pressure was measured 7 minutes after tracheal intubation.
Prediction power of the post-induction hypotension of carotid sonography and inferior vena cava sonography | 10 minutes after tracheal intubation
  To evaluate the ability of carotid sonography and inferior vena cava sonography for the post-induction hypotension in hypertensive patients undergoing general anesthesia, blood pressure was measured 10 minutes after tracheal intubation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea